CLINICAL TRIAL: NCT07207642
Title: Sweet Night (Musical Diffusion by Caregivers ): Effects of Musical Diffusion by Caregivers on Sleep Onset and Behavioral Regulation in a Protected Living
Acronym: Sweet nightMDC
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 25CH036; 2025-A00468-41 (Other: ANSM)
Record Dates: First submitted 2025-06-18; First posted 2025-10-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease or Associated Disorder
Keywords: Alzheimer's disease; Music intervention; Behavior disorder
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Passive EXPERIMENT: Measurement of the effects of a personalised music listening session at bedtime (play-list) for 10 days. Each patient is his or her own control. Behavioural and actigraphic data are collected and compared before, during and after the intervention.
  Interventions: Behavioral: Music intervention - passive listening
- Active EXPERIMENT: An intervention based on listening to audio books, led by a therapist for 10 evenings . Each patient is his or her own control and takes part in the entire experiment. Behavioural and actigraphic data are collected and compared before, during and after intervention.
  Interventions: Behavioral: Audio books intervention - active listening

INTERVENTIONS:
Behavioral: Music intervention - passive listening — Diffusion of familiar music in the bedrooms and living room before bedtime; passive and individual listening.
  Groups: Passive EXPERIMENT
Behavioral: Audio books intervention - active listening — Dynamic audio book listening, akin to active listening while respecting the rhythm of the evening . This type of listening involves concentrating specifically .
  Groups: Active EXPERIMENT

SUMMARY:
As the Alzheimer's disease progresses, caregivers and family members often focus on behavioral difficulties. In response to crises, immediate actions tend to favor restraints, either through medication or physical means. This work aims to improve the management of behavioral disturbances in patients with Alzheimer's disease through musical interventions (group or individual), particularly in advanced stages of the disease, where medical and family resources are insufficient. The investigators approach prioritizes NTM over medication as a mean to improve patient well-being. To this end, they have designed a study. The study focuses on creating a conducive environment for sleep by incorporating ritualized, familiar music sessions supervised by nursing staff after meals. To conduct this study, the actigraphy will be used to analyze participants' behavior both day and night, complemented by questionnaires and clinical observations.

ELIGIBILITY:
Inclusion Criteria:

* Non-opposition of the patient's legal guardian.
* Patients aged 60 and over, meeting the diagnostic criteria for Alzheimer's disease and related disorders.
* Patients living in a Protected Living Unit (PLU)
* If consuming psychotropic medications, they must have been stabilized for 3 months.
* If consuming level 2 or 3 analgesics, they must have been stabilized for 1 month.

Exclusion Criteria:

* Refusal to participate.
* Participation in a study on a drug /medical device / care technique that could affect sleep or behavior during the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 and over, meeting the diagnostic criteria for Alzheimer's disease and related disorders, living in a Protected Living Unit (PLU) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | Days 1 to 51
  Sleep duration will be measured by actigraphy (bracelet worn by the participants).

SECONDARY OUTCOMES:
Sleep onset and nocturnal awakenings reduction | Days 1 to 51
  Sleep onset latency and number of nocturnal awakenings measured by actigraphy.
Daytime agitation reduction | Days 1 to 51
  Cohen-Mansfield Agitation Inventory score, which assesses 29 items including: non-aggressive physical agitation (1-13), non-aggressive verbal agitation (14-17), physical agitation and aggression (18-26), and verbal agitation and aggression (27-29). A high score reflects intense agitation.
Mood improvement | Days 1 to 51
  Caregiver questionnaire: category scale : for agitation and mood.
Falls number reduction | Days 1 to 51
  Fall questionnaire include in the caregiver questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle ROUCH, Md, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France, France

IPD SHARING:
Plan to Share IPD: No